CLINICAL TRIAL: NCT06906198
Title: A Randomized, Double-Masked, Vehicle-Controlled, Single-Center Phase 1 Clinical Study Evaluating the Safety, Tolerability and Pharmacokinetics of 0.25%, 0.5% and 1.0% VVN461 Ophthalmic Solution
Brief Title: Pharmacokinetics of VVN461 Ophthalmic Solution
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VivaVision Biotech, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VVN461-CCS-101
Record Dates: First submitted 2024-12-03; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: dose-escalating
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- VVN461, 1.0% (Experimental): VVN461 Ophthalmic Solution, 1.0%
  Interventions: Drug: VVN461 Ophthalmic Solution 1.0%
- VVN461, 0.5% (Experimental): VVN461 Ophthalmic Solution, 0.5%
  Interventions: Drug: VVN461 Ophthalmic Solution 0.5%
- VVN461, 0.25% (Experimental): VVN461 Ophthalmic Solution, 0.25%
  Interventions: Drug: VVN461 Ophthalmic Solution 0.25%
- Vehicle (Placebo Comparator): VVN461 Ophthalmic Solution, Placebo
  Interventions: Drug: VVN461 Ophthalmic Solution Placebo

INTERVENTIONS:
Drug: VVN461 Ophthalmic Solution 1.0% — VVN461, 1.0%
  Arms: VVN461, 1.0%
Drug: VVN461 Ophthalmic Solution 0.5% — VVN461, 0.5%
  Arms: VVN461, 0.5%
Drug: VVN461 Ophthalmic Solution 0.25% — VVN461, 0.25%
  Arms: VVN461, 0.25%
Drug: VVN461 Ophthalmic Solution Placebo — Vehicle
  Arms: Vehicle

SUMMARY:
This is a single-center, double-masked, randomized, vehicle-controlled study conducted in China in adult healthy subjects

DETAILED DESCRIPTION:
This is a Phase I, randomized, double-masked, vehicle-controlled study to evaluate the safety, tolerability and pharmacokinetics of 0.25%, 0.5% and 1.0% VVN461 Ophthalmic Solution in healthy male and female volunteers in China.

The study consisted of a screening period (D-7 to D-1), a baseline visit (D-1), a single-dose period (D1), QID multi-dose period (D2 to D5), six times daily multi-dose period (D6 to D9), discharge (D10), and a follow-up/EOS (D16,+1D). During the single-dose period, subjects will receive one drop of VVN461 eye drops (0.25%, 0.5%, or 1.0%) or vehicle in the study eye. For the multi-dose period, subjects will receive one drop of VVN461 eye drop (0.25%, 0.5% or 1.0%) or vehicle in the study eye four or six times a day. PK blood samples will be collected before and after dosing at D1, D5 and D9.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 50 years at the time of signing the informed consent form.
* Males weighing ≥ 50.0kg and females ≥ 45.0kg; and with a body mass index (BMI = weight/height squared) of 19-26 kg/m2 (including thresholds).
* Best-corrected visual acuity (BCVA) ≥ 0.8 (standard logarithmic scale) in both eyes; intraocular pressure of 11-21 mmHg (including threshold) in both eyes; and slit-lamp examination of the anterior segment of the eye and funduscopic examination (funduscopic photographs) with no significant abnormality or an abnormality judged by the investigator to be not clinically significant.
* No clinically significant medical history of the liver, kidneys, gastrointestinal tract, nervous system, respiratory system (e.g., asthma, exercise-induced asthma, chronic obstructive pulmonary disease), hematological and lymphatic system, musculoskeletal system, rheumatological immunity, psychiatric abnormalities and metabolic abnormalities
* Physical examination, vital signs, 12-lead electrocardiogram and laboratory tests at screening are within normal values or the abnormalities are not clinically significant.

Exclusion Criteria:

* Known hypersensitivity or contraindications to the study drug or its components
* Anatomical anomalies in either eye
* History of eye surgery (other than blepharoplasty) or laser treatment of the eye (including keratoconus) in either eye
* Blepharoplasty on either eye within 3 months prior to screening
* History of subchoroidal or vitreous injection in either eye
* Infectious eye disease, immunological eye disease, inflammatory eye disease or ocular trauma in either eye within three months prior to screening;
* Use of topical ophthalmic medications (including artificial tears, proprietary drops and OTC ophthalmic medications) in either eye within 1 month prior to screening
* Using contact lens in either eye within 14 days prior to screening or unable to discontinue the use of contact lens during the study
* A history of eye disease such as glaucoma, corneal opacity, corneal degeneration, corneal dystrophy, uveitis, fundopathy, or other ophthalmic disease in either eye, which is assessed by the investigator to be contraindicated for participation in the trial.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Safety outcome | Baseline to Day 16
  Incidence of adverse events

SECONDARY OUTCOMES:
Time to maximum blood level | Maximum seen over Days 1 to 9
  Tmax
Area under the curve of blood levels until last observation | Integrated over Days 1 to 9
  AUC0-last
Area under the curve of blood levels extrapolated to infinity | Integrated over Days 1 to 9
  AUC0-inf
Half life of drug in blood | Integrated over Days 1 to 9
  t1/2

OTHER OUTCOMES:
Maximum concentration of drug in blood | Integrated over Days 1 to 9
  Cmax

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China